CLINICAL TRIAL: NCT05930028
Title: A Randomized, Double-blind, Multi-center, Phase III Trial to Evaluate the Efficacy and Safety of BR1017A and BR1017B Combination Therapy in Essential Hypertension Patients With Primary Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of BR1017A and BR1017B Combination Therapy in Essential Hypertension Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FAEC-CT-301
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Essential Hypertension; Primary Hypercholesterolemia
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fimasartan/Ezetimibe/Atorvastatin (Experimental): BR1017A+BR1017B(Experimental Group)
  Interventions: Drug: Fimasartan; Drug: Ezetimibe/Atorvastatin
- Fimasartan (Active Comparator): BR1017A(Control Group 2)
  Interventions: Drug: Fimasartan; Drug: Ezetimibe/Atorvastatin Placebo
- Ezetimibe/Atorvastatin (Active Comparator): BR1017B(Control Group 1)
  Interventions: Drug: Ezetimibe/Atorvastatin; Drug: Fimasartan Placebo

INTERVENTIONS:
Drug: Fimasartan — Subjects take the investigational products once a day for 8 weeks.
  Other Names: BR1017A
  Arms: Fimasartan; Fimasartan/Ezetimibe/Atorvastatin
Drug: Ezetimibe/Atorvastatin — Subjects take the investigational products once a day for 8 weeks.
  Other Names: BR1017B
  Arms: Ezetimibe/Atorvastatin; Fimasartan/Ezetimibe/Atorvastatin
Drug: Fimasartan Placebo — Subjects take the investigational products once a day for 8 weeks.
  Other Names: BR1017A-1
  Arms: Ezetimibe/Atorvastatin
Drug: Ezetimibe/Atorvastatin Placebo — Subjects take the investigational products once a day for 8 weeks.
  Other Names: BR1017B-1
  Arms: Fimasartan

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety by comparing BR1017A+BR1017B treatment group to BR1017A treatment group and BR1017B treatment group respectively at Week 8 in essential hypertension patients with primary hypercholesterolemia

ELIGIBILITY:
<Inclusion Criteria>

Screening

* Patients with essential hypertension and primary hypercholesterolemia
* If patients are being treated with antihypertensive/antihyperlipidemic drugs at screening (V1), they should be determined to be medically reasonable by investigator about discontinuing existing antihypertensive/ antihyperlipidemic drugs during the clinical trial
* Patients who have an fasting triglyceride (TG) < 400 mg/dL and LDL-C ≤ 250 mg/dL at Screening (V1)
* Voluntarily provided a written consent to participate in this clinical study
* Able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion

Randomization

* Patients who meet the following criteria of blood pressure measured in selected reference arm before randomization at baseline(V3)

  * 140 mmHg ≤ MSSBP < 180 mmHg
  * MSDBP < 110 mmHg
* Patients who meet the criteria of fasting serum lipid levels and risk factors at pre-baseline (V2) after undergoing the therapeutic lifestyle change (TLC)
* Patients who have an fasting triglyceride (TG) < 400 mg/dL and LDL-C ≤ 250 mg/dL after undergoing the therapeutic lifestyle change (TLC) for at least 4 weeks before pre-baseline (V2)

<Exclusion Criteria>

* Patients with blood pressure results showing MSSBP ≥ 180 mmHg or MSDBP ≥ 110 mmHg in the selected reference arm at screening(V1) or Baseline(V3)
* Patients with a difference of MSSBP ≥ 20 mmHg and MSDBP ≥ 10 mmHg in blood pressure measured three times on both arms at screening(V1)
* Patients with past history and comorbidities at screening(V1) under the following criteria:

  * Patients with secondary hypertension: Secondary hypertension is not limited to the following diseases; (e.g., coarctation of the aorta, hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma and polycystic kidney disease, etc.)
  * Patients with secondary hyperlipidemia: Secondary hyperlipidemia is not limited to the following diseases; (e.g., Chronic renal failure, nephrotic syndrome, obstructive liver disease, hypothyroidism, dysproteinemia, etc.)
  * Patients with orthostatic hypotension accompanied by symptoms

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Mean sitting systolic blood pressure | 8weeks from Baseline Visit
  The change of mean sitting systolic blood pressure from baseline in BR1017A+BR1017B at Week 8 compared to BR1017B
LDL-C | 8weeks from Baseline Visit
  The percent of change in LDL-C from baseline in BR1017A+BR1017B at Week 8 compared to BR1017A

SECONDARY OUTCOMES:
LDL-C | 8weeks from Baseline Visit
  The percent of change in LDL-C from baseline in BR1017A+BR1017B at Week 8 compared to BR1017B
Mean sitting systolic blood pressure | 8weeks from Baseline Visit
  The change of mean sitting systolic blood pressure from baseline in BR1017A+BR1017B at Week 8 compared to BR1017A

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No